CLINICAL TRIAL: NCT07222410
Title: Closed Loop Oxygen Control in COPD Patients Treated With Nasal High Flow in the Hospital
Brief Title: Closed Loop Oxygen Control in Chronic Obstructive Pulmonary Disease (COPD) Patients Treated With Nasal High Flow in the Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIA-334
Record Dates: First submitted 2025-10-23; First posted 2025-10-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: COPD
Keywords: COPD; closed loop oxygen control; hypoxemia; nasal high flow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Airvo 3 (with OptiO2) OptiO2 mode on (Experimental)
  Interventions: Device: Closed loop oxygen control
- Airvo 3 (with OptiO2) OptiO2 mode off (Active Comparator)
  Interventions: Device: Manual titration

INTERVENTIONS:
Device: Closed loop oxygen control — Nasal high flow with closed loop oxygen control
  Arms: Airvo 3 (with OptiO2) OptiO2 mode on
Device: Manual titration — Nasal high flow with manual titration
  Arms: Airvo 3 (with OptiO2) OptiO2 mode off

SUMMARY:
The trial aims to evaluate whether the Airvo 3 device in OptiO2 mode can maintain patients' SpO2 levels within the target range better than manual oxygen titration in hospitalized COPD patients with hypoxemia/respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Has cognitive ability to provide informed consent
* Aged 22 years or older
* Hospitalized with hypoxemia/respiratory distress
* Diagnosis of COPD
* Candidate for/currently prescribed nasal high flow (flow rate of at least 25 L/min) with supplemental oxygen, as assessed by the investigator
* Expected duration of oxygen and nasal high flow therapy >24 hours (not necessarily continuous)

Exclusion Criteria:

* Receiving Non Invasive Ventilation (NIV) or indicated for NIV as per European Respiratory Society /American Thoracic Society guidelines
* Hemodynamic instability (systolic blood pressure <90mmHg or requirement for vasopressor or inotropic support)
* Patient receiving end of life care
* Nasal or facial conditions precluding use of nasal high flow
* Pregnancy or breastfeeding
* Cognitive impairment or impaired consciousness precluding informed consent
* Unsuitable for adhesive finger pulse oximetry, as assessed by the investigator
* Any other condition which, at the investigator's discretion, is believed to present a safety risk to the patient if included
* The presence of any active comorbidities that affect the patient's condition importantly in the next 30 days, as assessed by the investigator
* Has already participated in this clinical trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of time with SpO2 in target range over period of observation | 24 hours
Percentage of time with SpO2 out of target range over period of observation | 24 hours

SECONDARY OUTCOMES:
Count of number of adjustments in FiO2 by clinical staff over observation period | 24 hours
Percentage of time with SpO2 above target range over period of observation | 24 hours
Percentage of time with SpO2 below target range over period of observation | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Sensitivity of data, data will be used for FDA submission